CLINICAL TRIAL: NCT01192321
Title: Visual Outcomes After Bilateral Surgical Cataract Phacoemulsification: AcrySof Toric Intraocular Lens (IOL) Implantation Compared to Monofocal IOL Implantation
Brief Title: Visual Outcomes After Bilateral Surgical Cataract Phacoemulsification: AcrySof Toric IOL Implantation Compared to Monofocal IOL Implantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision to close study based on low enrollment
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M09-047
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Cataract
Keywords: intraocular lens; Toric
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toric T3 - T9 (Experimental): Bilateral implantation of a Toric intraocular lens (IOL) models T3, T4, T5, T6, T7, T8 or T9
  Interventions: Device: Toric T3 - T9
- Monofocal (Active Comparator): Bilateral implantation of a monofocal intraocular lens (IOL) model with no toric component.
  Interventions: Device: Monofocal

INTERVENTIONS:
Device: Toric T3 - T9 — Bilateral implantation of Alcon AcrySof Toric Intraocular Lens (IOL) models SN60T3 through SN60T9 following cataract removal.
  Arms: Toric T3 - T9
Device: Monofocal — Bilateral implantation of any monofocal Intraocular Lens (IOL) following cataract removal.
  Arms: Monofocal

SUMMARY:
The objectives of this study are to assess and compare bilateral uncorrected distance visual acuity and distance spectacle independence post bilateral implantation of AcrySof Toric Intraocular Lenses (IOLs) and monofocal IOLs. Secondary outcomes will include cost of eyeglass purchased and patient vision-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* are willing and able to understand and sign an informed consent;
* are willing and able to attend postoperative examinations per protocol schedule;
* are ≥ 21 years of age, of either gender and any race;
* have bilateral, age related, cataracts;
* have planned cataract removal via phacoemulsification with implantation of an intraocular lens (IOL);
* are available to undergo second eye surgery within 6 weeks of the first eye surgery;
* are in good ocular health, with the exception of cataracts;
* are free of disease(s)/condition(s) listed in the "Precautions" section of the AcrySof Toric and monofocal package inserts: choroidal hemorrhage, chronic severe uveitis, concomitant severe eye disease, extremely shallow anterior chamber, medically uncontrolled glaucoma, microphthalmos, non-age-related cataract, proliferative diabetic retinopathy (severe), severe corneal dystrophy, severe optic nerve atrophy, irregular corneal astigmatism and color vision deficiencies.
* have regular corneal astigmatism;
* qualify for bilateral AcrySof Toric IOLs on the AcrySof Toric Calculator (www.acrysoftoriccalculator.com)
* are able to obtain pupil dilation ≥ 5.0 mm
* are able to read and understand one of the following languages: Dutch, French, German

Exclusion Criteria:

* previous corneal surgery and/or reshaping
* abnormality, disease and/or conditions of the cornea (i.e. keratoconus, corneal dystrophy, keratitis, corneal scar, etc.), which would clinically contra-indicate the implantation of a toric intraocular lens
* planned multiple procedures during cataract/IOL implantation surgery
* planned limbal relaxing incision (LRI), Excimer laser treatment or similar procedure prior to or during the course of the study
* an ocular disease and/or condition that may compromise visual acuity levels (i.e. glaucoma, diabetic retinopathy, amblyopia, etc.)
* pregnant, lactating or planning pregnancy during course of study. Subjects who become pregnant during the study will not be discontinued; however, data may be excluded from the effectiveness analyses because pregnancy can alter refraction and visual acuity results. Data will be collected on the CRF as observations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Uncorrected Distance Visual Acuity | 6 Months After Surgery
  Visual Acuity (VA) is measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Spectacle Independence | 6 Months After Surgery
  Spectacle Independence (the ability of the patient to go without corrective lenses) measured by a subjective patient questionnaire.

SECONDARY OUTCOMES:
Vision-related Quality of Life | 6 Months After Surgery
  Vision related quality of life as measured by a subjective subject questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Paris, France